CLINICAL TRIAL: NCT06381362
Title: Italian Registry of Minimally Invasive Pancreatic Surgery (IGOMIPS)
Brief Title: Italian Registry of Minimally Invasive Pancreatic Surgery
Acronym: IGOMIPS
Status: Recruiting | Type: Observational
Sponsor: Associazione Italiana per lo Studio del Pancreas (Other)
Responsible Party: Sponsor
Other Study IDs: IGOMIPS
Record Dates: First submitted 2024-03-13; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Minimally invasive pancreatic surgery — Minimally invasive pancreatic surgery

SUMMARY:
Assess the prevalence of minimally invasive pancreatic surgery in the country and its outcomes

DETAILED DESCRIPTION:
Since 1994, when the first pancreatectomy surgeries, distal and proximal, conducted minimally invasively, were published, efforts have been made to understand the value of this approach in the context of a surgery as complex and burdened with specific complications as pancreatic surgery. The adoption of such an approach with regard to pancreatic surgery has been less rapid and parceled out than in other surgical fields and not supported by a large body of scientific publications. However, worldwide, referral centers for pancreatic surgery routinely use the minimally invasive approach in selected cases, and its diffusion has recently shown a marked increase. Even in Italy, a recent survey promoted by some of the major surgical societies showed a fair diffusion of the use of the minimally invasive approach in pancreatic surgery but with extremely variable ways and uses in the different territorial realities with evident and potentially risky paradoxes. Monitoring the diffusion of minimally invasive pancreatic surgery, the methods of application and the results of this approach has become of primary importance and for this reason the foundation of a national registry has been proposed by several scientific surgical societies.

This study aims to investigate what is the real diffusion of minimally invasive techniques in Italy and what postoperative outcomes the adoption of this approach generates.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Underwent minimally invasive pancreatic surgery

Exclusion Criteria:

* Pregnant woman
* Minor or unable to give informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will involve all patients undergoing at participating centers a pancreatic surgery performed by minimally invasive technique (e.g., laparoscopic, robotic), over the age of 18 years, capable of expressing consent to the study.
Sampling Method: Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Postoperative short-term outcomes | 90 days
  any complication graded according to Clavien-Dindo classification
Long-term oncological outcomes | 2 years
  Disease recurrence or disease related death

SECONDARY OUTCOMES:
Rate of cases that after a minimally invasive approach had to be converted to and open approach | Intraoperative
  Intraoperative conversion to open surgery for any reason
Surgeon learning curve | Intraoperative
  Variation of surgical time according to the registered case-load as operating surgeon and first assistant
Surgeon learning curve | Intraoperative
  Variation of intraoperative blood-loss according to the registered case-load as operating surgeon and first assistant
Surgeon learning curve | Intraoperative
  Variation of intraoperative complications rate according to the registered case-load as operating surgeon and first assistant
Surgeon learning curve | Intraoperative
  Variation of conversion rate according to the registered case-load as operating surgeon and first assistant

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Zerbi, Prof., Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Giovanni Capretti, Milan, Italy

IPD SHARING:
Plan to Share IPD: No